CLINICAL TRIAL: NCT00836160
Title: Comparing Efficacy Between Anti-microtubule and Non-anti-microtubule as 3th Therapy After 2nd Line EGFR-TKI Therapy
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OTW-DUM-2008/1
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Cancer
Keywords: EGFR-TKI therapy; NSCLC; Efficacy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
This is an observational prospective study that investigates only daily practice. The prescription of anti-cancer medicine is separated from the decision to include the patient in this study. In addition, the assignment of the patient to a particular therapy or therapeutic strategy is not decided in advance by this study protocol, but falls within current practice.

The patient who fulfils eligible criteria will be enrolled when starts to receive the second-line EGFR-TKI therapy. The frequency of tumor response evaluation by RECIST criteria follows the investigator's discretion as daily practice.

ELIGIBILITY:
Inclusion Criteria:

* At least one measurable lesion according to RECIST criteria
* Histologically or cytologically confirmed NSCLC of adeno histology
* Locally progressed or metastasized on or after first-line chemotherapy. The imaging evidence of disease progression can be either chest X ray, CT or MRI assessment on measurable lesions. If no measurable lesion is available, evaluable lesions are acce

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The EGFR-TKI receiver who are suitable for third-line therapy will be followed up for the regimen of the third-line anti-microtubule agents or non-anti-microtubule agents
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
PFS of the third-line therapy | 9 months

SECONDARY OUTCOMES:
Overall objective tumor response (complete response [CR] + partial response [PR]) of the third-line therapy by RECIST criteria | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Gueishan Township, Taiwan